CLINICAL TRIAL: NCT00324363
Title: Safety and Efficacy of Exenatide in Patients With Type 2 Diabetes Using Metformin or Sulfonylureas and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-MC-GWBA
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; diabetes; Amylin; Lilly; China
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Placebo lead-in; exenatide 5 mcg for 4 weeks; exenatide 10 mcg for 12 weeks
  Interventions: Drug: exenatide
- Placebo (Placebo Comparator): Placebo in volume equal to exenatide
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day for 16 weeks
  Other Names: Byetta
  Arms: Exenatide
Drug: Placebo — subcutaneous injection twice daily in volumes equal to exenatide
  Arms: Placebo

SUMMARY:
This study is designed to compare the effects of twice-daily exenatide plus oral antidiabetic (OAD) agents and twice-daily placebo plus OAD with respect to glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Treated with a stable dose of one of the following for at least 3 months prior to screening: * >=1000 mg/day immediate-release metformin; or metformin >=1000 mg/day and sulfonylurea; or sulfonylurea/metformin combination therapy.
* HbA1c between 7.1% and 11.0%, inclusive.
* Body Mass Index (BMI) >21 kg/m^2 and <35 kg/m^2.

Exclusion Criteria:

* Have participated in this study previously, or any other study using exenatide or GLP-1 analogs.
* Have participated in an interventional, medical, surgical, or pharmaceutical study within 30 days of screening.
* Have characteristics contraindicating metformin or sulfonylurea use.
* Have been treated with exogenous insulin for more than 1 week within the 3 months prior to screening.
* Have used drugs for weight loss within 1 month of screening.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that exenatide (before morning and evening meals) produces a greater decrease in HbA1c than placebo in patients with type 2 diabetes and inadequate glycemic control taking metformin alone or metformin and sulfonylureas. | 16 weeks

SECONDARY OUTCOMES:
To compare exenatide and placebo groups with respect to: *safety and tolerability; *proportion of patients achieving HbA1c<=7%; *body weight; *incidence and rate of hypoglycemic events; *glucose measurements | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (14):
- China (5):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Sichuan
- India (3):
  - Research Site, Chennai
  - Research Site, Mumbai
  - Research Site, Pune
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Sungnam City
- Taiwan (4):
  - Research Site, Chiayi City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei

REFERENCES:
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] Gao Y, Yoon KH, Chuang LM, Mohan V, Ning G, Shah S, Jang HC, Wu TJ, Johns D, Northrup J, Brodows R. Efficacy and safety of exenatide in patients of Asian descent with type 2 diabetes inadequately controlled with metformin or metformin and a sulphonylurea. Diabetes Res Clin Pract. 2009 Jan;83(1):69-76. doi: 10.1016/j.diabres.2008.09.037. Epub 2008 Nov 18. PMID 19019476